CLINICAL TRIAL: NCT00629239
Title: A 4-week Double-blind, Placebo-controlled, Randomized, Parallel Group Phase IIa Study to Assess the Tolerability/Safety and Efficacy of Inhaled AZD4818 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tolerability/Safety and Efficacy of Inhaled AZD4818 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: TOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Bengt Larsson/MD PhD Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3540C00005
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; tolerability; inhalation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — AZD-4818

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD4818
  Interventions: Drug: AZD4818
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4818 — Dry Powder, inhalation, b.i.d., 4 weeks
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to see if treatment with AZD4818 for four weeks is tolerable, safe and effective in treating COPD and, if so, how it compares with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, with symptoms for more than 1 year
* Current or ex-smokers with a smoking history of at least 10 pack-years (1 pack-year=20 cigarettes/day for 1 year)
* Lung function (FEV1) 40 to 80% of the predicted normal value after using a short acting bronchodilator

Exclusion Criteria:

* Clinical suspicion of active tuberculosis
* Any current clinically significant respiratory tract disorder other than COPD
* History of current clinically relevant arrhythmia, heart block, ECG abnormalities, or unstable angina

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huib AM Kerstjens, MD, PhD, Principal Investigator — University Medical Centre, Groningen, The Netherlands
Locations (12):
- Denmark (3):
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense C
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Preitilä
  - Research Site, Tampere
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Groningen
- Norway (3):
  - Research Site, Elverum
  - Research Site, Oslo
  - Research Site, Trondheim
- Research Site, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was excluded in the analysis sets since this participat is non-informative both in terms of efficacy and safety, and was immediately withdrawn for non-treatment related reasons. AZD4818 Turbuhaler group will include 33 patients in all other sections
Groups:
- AZD4818: AZD4818 Turbuhaler
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD4818 | Placebo
Started | 34 | 32
Completed | 26 | 28
Not Completed | 8 | 4
Not completed — Adverse Event | 7 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD4818 | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age Continuous [Mean (Full Range); unit: years] | 65 [51 to 78] | 66 [42 to 77] | 65 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Adverse Events
Description: Number of patients who had an Adverse Event
Time Frame: At all study visits
Measure: Number; unit: Participants
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 22 | 27

2. Secondary Outcome: Forced Expiratory Volume 1 (FEV1)
Description: Change in (FEV1) from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L | -0.083 (-0.5) [-0.5 to 0.62] | -0.149 (-1.05) [-1.05 to 0.22]

3. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Change in FVC from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L | -0.044 (-1.02) [-1.02 to 0.950] | -0.240 (-1.54) [-1.54 to 0.730]

4. Secondary Outcome: Vital Capacity (VC)
Description: Change in VC from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 32 | 32
L | -0.022 (-0.86) [-0.86 to 1.92] | -0.022 (-1.25) [-1.25 to 0.860]

5. Secondary Outcome: Inspiratory Capacity (IC)
Description: Change from IC baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: L
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L | -0.117 (-1.02) [-1.02 to 0.83] | -0.038 (-0.73) [-0.73 to 1.04]

6. Secondary Outcome: Forced Expiratory Flow (FEF) 25%-75%
Description: Change in FEF from baseline to end of treatment
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: L/s
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L/s | -0.027 (-0.19) [-0.19 to 0.18] | 0.006 (-0.49) [-0.49 to 0.51]

7. Secondary Outcome: Peak Expiratory Flow (PEF) Morning
Description: Change from average during run-in to average during treatment
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L/min | -9.10 (-62.8) [-62.8 to 45.9] | -4.47 (-43.3) [-43.3 to 32.9]

8. Secondary Outcome: Peak Expiratory Flow (PEF) Evening
Description: Change in PEF from average during run-in to average during treatment
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
L/min | -12.4 [-42.9 to 35.9] | -1.90 [-33.0 to 34.2]

9. Secondary Outcome: The Clinical COPD ( Chronic Obstructive Pulmonary Disease) Questionnaire (CCQ) Total
Description: Change from baseline to end of treatment in score , The total scores vary between 0 (never/not limited at all) to 6 (almost all the time/totally limited)
Time Frame: Before treatment and after 1, 2, 3 and 4 weeks of treatment
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Score on a scale | 0.250 (-1.08) [-1.08 to 2.0] | 0.044 (-1.58) [-1.58 to 3.08]

10. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Breathlessness
Description: Change from average during run-in to average during treatment. Scores on a Scale, 5-point Likert-type scale, ranging from 0 (none) to 4 (severe).
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Scores on a scale | 0.159 (-0.446) [-0.446 to 1.23] | -0.007 (-1.18) [-1.18 to 1.40]

11. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Chest Tightness
Description: as for outcome 10
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Score on a scale | 0.170 (-0.823) [-0.823 to 2.44] | 0.024 (-0.807) [-0.807 to 0.847]

12. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Cough Score
Description: as for outcome 10
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Scores on a scale | 0.064 (-0.431) [-0.431 to 1.15] | -0.103 (-1.91) [-1.91 to 0.867]

13. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Symptoms, Sleep Score
Description: Change from average during run-in to average during treatmentScores on a Scale, 5-point Likert-type scale, ranging from 0 (none) to 4 (severe).
Time Frame: Daily during run-in and treatment
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
Scores on a scale | 0.085 [-0.926 to 1.15] | 0.000 [-1.19 to 0.889]

14. Secondary Outcome: 6-minute Walk Test
Description: Change from baseline to end of treatment
Time Frame: Before treatment and after 4 weeks of treatment
Measure: Mean (Full Range); unit: meter
Arm/Group | AZD4818 | Placebo
Number analyzed (Participants) | 33 | 32
meter | -8.67 (-163) [-163 to 90] | -6.67 (-125) [-125 to 112]

ADVERSE EVENTS:
Arm/Group | AZD4818 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/32
Other Adverse Events (participants affected / at risk) | 22/33 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4818 (N=33) | Placebo (N=32)
Deep Venous Thrombosis Left Lower Leg (Vascular disorders) | 1 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4818 (N=33) | Placebo (N=32)
Chronic obstructuve pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7
nasopharyngitis (Infections and infestations) | 1 | 8
Tremor (Nervous system disorders) | 5 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate with AZ in regard to the contents and formation of any publication or disclosure and to considerate the comments,views and opinions offered by AZ. Prior to any publication or disclosure the PI will provide AZ with preliminary data and drafts of proposed publication or disclosure and the proposed final manuscript. AZ will have a period of 30 days from receipt of the proposed final manuscript to review and may require submission for publication or disclosure be delayed